CLINICAL TRIAL: NCT01482039
Title: Patient Attitudes Regarding Abdominal Versus Transvaginal Ultrasonography for Assessment of the Cervical Length in Low Risk Patients: a Randomized Trial
Brief Title: Patient Attitudes Toward Ultrasound Measurement of Cervical Length
Acronym: TVUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Women and Children's Research (Other)
Responsible Party: Principal Investigator, Stephanie T. Romero, Principal Investigator, Intermountain Women and Children's Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Sonographic Cervical Length
Record Dates: First submitted 2011-11-25; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Cervical Insufficiency
Keywords: short cervix; cervical shortening; preterm birth
MeSH Terms: conditions — Uterine Cervical Incompetence; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Ultrasound (No Intervention): Current standard of care - one abdominal view of the cervix to rule out placenta previa
- Sequential Screen (Experimental): Start with 3 abdominal views of the cervix with measurement. If 3 adequate views cannot be obtained, or if measurement is less than 3cm, then will perform transvaginal scan for measurement.
  Interventions: Procedure: Sequential ultrasound
- Screening Transvaginal Ultrasound (Experimental): Obtain 3 adequate cervical length measurements using transvaginal ultrasound
  Interventions: Procedure: Transvaginal ultrasound

INTERVENTIONS:
Procedure: Sequential ultrasound — Abdominal ultrasound first; obtain 3 adequate measurements. If 3 adequate views not obtained or if measurement less than 3 cm, perform transvaginal ultrasound for measurement.
  Arms: Sequential Screen
Procedure: Transvaginal ultrasound — Obtain 3 transvaginal ultrasound cervical length measurements
  Arms: Screening Transvaginal Ultrasound

SUMMARY:
The investigators propose a prospective evaluation of methods to assess cervical length for uncomplicated singleton gestations between 18-28 weeks presenting to the MFM office for routine mid pregnancy ultrasound. The investigators hypothesize that a sequential approach to screening of the cervix (which consists of initial transabdominal evaluation first with transvaginal ultrasound reserved only for those patients in whom the cervix appears short on transabdominal exam or when adequate views cannot be obtained with the transabdominal approach alone) will take less time, will result in the same number of adequate views of the cervix and will have higher patient satisfaction that a universal transvaginal screening approach.

OBJECTIVE

To determine the best strategy for cervical length screening in uncomplicated singleton gestations between the gestational ages of 18-28 weeks.

Primary outcome:

1) Time required to obtain adequate views of the cervical length.

Secondary outcomes:

1. Patient satisfaction with ultrasound experience as measured by patient questionnaire
2. Number of adequate views of the cervix obtained with each approach

STUDY DESIGN

This is a prospective study to compare strategies for cervical length measurements in uncomplicated singleton gestations seen in the MFM office for routine mid pregnancy fetal well being ultrasound between 18-28 weeks gestation. The different strategies include 1) Transabdominal assessment of the cervix (current standard), 2) Sequential evaluation of the cervical length (transabdominal followed by transvaginal if necessary due to short cervix or inadequate transabdominal views), and 3) Transvaginal cervical length assessment. Patients with an uncomplicated singleton gestation presenting for a routine mid pregnancy ultrasound between 18-28 weeks will be randomized into one of the three groups noted above after consent is obtained. Ultrasound examination will then take place and data collected. The various strategies listed above will be compared for the following:

1. Time required to obtain views of the cervix

   1. Time from initiation of exam to completion of cervical assessment
   2. Time for completion of entire exam
2. Patient satisfaction

   1. Comfort/Discomfort of exam procedure
   2. Overall impression of exam process
3. Number of adequate views of the cervix obtained

Maternal demographics including age, parity, weight, height and due date/gestational age will also be obtained for all consenting patients.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

Preterm birth is a significant problem in the United States and worldwide. Approximately twelve percent of births in the US occur before 37 weeks and are considered preterm. Of these, 80% are considered "spontaneous preterm deliveries" (as opposed to iatrogenic) and are related to preterm labor or preterm rupture of membranes (Arias, 2003). Certain pregnancy characteristics have been identified to determine those patients at risk for preterm delivery. These include a history of preterm birth (Esplin, 2008), uterine anomalies, multiple gestation, among other things, both modifiable and not (Gardosi, 2000; Ananth, 2006). However, an important risk factor that can be identified is the presence of specific changes in the cervix, such as cervical shortening, and in fact, studies indicate that the risk of spontaneous preterm birth increases as cervical length decreases (Iams, 1996; Hibbard, 2000).

Some authors now advocate the universal screening of all pregnant women for cervical shortening at the time of the ultrasound that is performed at 18-28 weeks in most women. However, the best approach to evaluate the cervix in low risk patients (those without an identifiable risk factor) remains controversial.

PROTOCOL

1. Patients will be identified in the Maternal Fetal Medicine office and consented for randomization at the time of presentation for previously scheduled mid-trimester ultrasound
2. Patients will be given randomly generated treatment allocations within sealed opaque envelopes. Once a patient has consented to enter the trial, the envelope will be opened by the ultrasonographer to determine the assigned treatment regimen.
3. Patients will be randomized into one of three groups:

   1. Standard US evaluation
   2. Sequential US evaluation
   3. Transvaginal cervical length screening
4. Maternal demographics including maternal age, height, weight, parity, and gestational age will be collected from the patient as part of the patient questionnaire. Ultrasound exam data including measurements of the fetal biometry, presence of fetal anomalies, placental location and amniotic fluid volume will be collected from the official ultrasound report.

   1. Patients will be assigned a unique study ID number at the time of enrollment and all information including time of ultrasound procedures, clinical data and adequacy of cervical measurement will be linked by the ID number
   2. All data will be entered into an electronic data base in a de-identified fashion and kept in a secure, encrypted web-based database management program (RedCap).

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* between 18-28 weeks

Exclusion Criteria:

* presence of cerclage
* known short cervix
* prior preterm birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Time | Assessed on the day of ultrasound (one single visit)
  The time it takes to perform the assessment of the cervix will be recorded, as well as the time it takes to perform the entire exam.

SECONDARY OUTCOMES:
Patient satisfaction | Assessed the day of the ultrasound (one single visit)
  Participants will complete a survey indicating their opinions about the ultrasound experience.
Ultrasound adequacy | Assessed on the day of the ultrasound (one single visit)
  Assess the frequency with which adequate views of the cervix can be obtained using transabdominal vs transvaginal ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Romero, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Esplin MS, O'Brien E, Fraser A, Kerber RA, Clark E, Simonsen SE, Holmgren C, Mineau GP, Varner MW. Estimating recurrence of spontaneous preterm delivery. Obstet Gynecol. 2008 Sep;112(3):516-23. doi: 10.1097/AOG.0b013e318184181a. PMID 18757647
- [Background] Adams MM, Elam-Evans LD, Wilson HG, Gilbertz DA. Rates of and factors associated with recurrence of preterm delivery. JAMA. 2000 Mar 22-29;283(12):1591-6. doi: 10.1001/jama.283.12.1591. PMID 10735396
- [Background] Iams JD, Goldenberg RL, Meis PJ, Mercer BM, Moawad A, Das A, Thom E, McNellis D, Copper RL, Johnson F, Roberts JM. The length of the cervix and the risk of spontaneous premature delivery. National Institute of Child Health and Human Development Maternal Fetal Medicine Unit Network. N Engl J Med. 1996 Feb 29;334(9):567-72. doi: 10.1056/NEJM199602293340904. PMID 8569824
- [Background] Hibbard JU, Tart M, Moawad AH. Cervical length at 16-22 weeks' gestation and risk for preterm delivery. Obstet Gynecol. 2000 Dec;96(6):972-8. doi: 10.1016/s0029-7844(00)01074-7. PMID 11084188
- [Background] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Background] Fonseca EB, Celik E, Parra M, Singh M, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Progesterone and the risk of preterm birth among women with a short cervix. N Engl J Med. 2007 Aug 2;357(5):462-9. doi: 10.1056/NEJMoa067815. PMID 17671254
- [Background] Stone PR, Chan EH, McCowan LM, Taylor RS, Mitchell JM; SCOPE Consortium. Transabdominal scanning of the cervix at the 20-week morphology scan: comparison with transvaginal cervical measurements in a healthy nulliparous population. Aust N Z J Obstet Gynaecol. 2010 Dec;50(6):523-7. doi: 10.1111/j.1479-828X.2010.01225.x. Epub 2010 Sep 16. PMID 21133862